CLINICAL TRIAL: NCT04553848
Title: Augmented Reality and Treadmill Training After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director of Research and Evaluation, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1606744
Record Dates: First submitted 2020-09-03; First posted 2020-09-18 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Augmented Reality+ Treadmill training (Experimental): Participants allocated to this group will receive treadmill training with body weight support (BWS) incorporating augmented feedback games chosen to address clinically perceived deficits using the C-Mill training system.
  Interventions: Behavioral: Augmented Reality; Behavioral: Treadmill training
- Treadmill training (Active Comparator): Participants allocated to this group will receive treadmill training with body weight support (BWS) using the C-Mill training system.
  Interventions: Behavioral: Treadmill training
- Over ground training/standard of care (Active Comparator): Participants allocated to this group will receive over ground balance and mobility training that would be considered standard of care in outpatient rehabilitation.
  Interventions: Behavioral: Over ground training/standard of care

INTERVENTIONS:
Behavioral: Augmented Reality — Augmented Reality (AR) systems are computer-based applications that allow an individual to view a simulated environment and dynamically interact within this environment in real-time. Augmented reality activities will be chosen by the therapist based on the primary deficits assessed during baseline testing.
  Arms: Augmented Reality+ Treadmill training
Behavioral: Treadmill training — The goal of each session will be to increase balance and mobility challenge by increasing speed and minimizing BWS. Appropriate BWS will be chosen at the beginning of each training session. Participants will walk for 1 minute on the treadmill at 30%, 20% and 10% BWS. Maximum walking speed will be determined at each level of BWS and the participant will spend the remainder of the session ambulating with BWS at which they were able to achieve maximum walking speed. Additional BWS will be provided up to 30% of the participant's total body weight if the treating therapist identifies safety concerns or unfavorable gait kinematics. If a safe and kinematically appropriate gait pattern is unable to be achieved at up to 30% BWS, the previously determined walking speed will be reduced to achieve a safe and appropriate walking pattern. Participants will be encouraged not to use upper extremity support while ambulating with BWS.
  Arms: Augmented Reality+ Treadmill training; Treadmill training
Behavioral: Over ground training/standard of care — Standard of care interventions to address balance and mobility deficits will be chosen from a list of commonly used interventions in outpatient therapy. The goal of each session will be to increase balance and mobility challenge in an over ground condition focusing treatment in the following areas:
  * Biomechanical Constraints
  * Stability Limits
  * Anticipatory Postural Adjustments
  * Reactive Postural Response
  * Sensory Orientation
  * Stability in Gait
  Arms: Over ground training/standard of care

SUMMARY:
Up to 40 participants will be enrolled in this study in order to obtain complete data on 30 participants. The investigators will be assessing if Augmented reality in combination with treadmill training is safe and feasible to use in the clinical environment with participants who have chronic TBI and if there is a signal of effect that this intervention may be more beneficial than treadmill training alone or standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a TBI requiring inpatient rehabilitation
* > 1 year post TBI
* 18-65 years of age
* Not currently participating in any other research study to address balance and gait impairment
* Not currently participating in physical therapy
* Ambulates with minimal assistance and/or assistive device
* Self-report of ongoing balance deficits and mobility deficits
* Score of 75 or below on CB&M
* No history of other neurological disorders affecting balance
* No seizures within the last year
* No history of psychiatric disorder requiring hospitalization
* Ability to follow directions and complete standardized instructions

Exclusion Criteria:

- No pregnant or lactating females (Potential female participants will be informed that risks to pregnant or lactating females are unknown; then they will be asked if they are pregnant or lactating, or if they could be pregnant. If there is any uncertainty, they will not be included in the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Community Balance and Mobility Scale | Baseline to Week 8
  13 activities scored from 0-96, higher numbers reflect greater balance

SECONDARY OUTCOMES:
10 meter walk test | Baseline, Week 4, and Week 8
  total time to walk 10 meters
6 minute walk test | Baseline, Week 4, and Week 8
  distance walked in 6 minutes
Timed Up and Go | Baseline, Week 4, and Week 8
  received verbal instructions to stand up from chair, walk 3 meters, cross a line marked on the floor, turn around, walk back and sit down
Timed Up and Go Cognitive Test | Baseline, Week 4, and Week8
  receive verbal instructions to stand up from a chair, walk 3 meters, cross a line marked on the floor, turn around, walk back and sit down while counting backward by threes from a randomly selected number between 20 and 100
Timed Up and Go Manual | Baseline, Week 4, and Week 8
  receive verbal instructions to stand up from a chair, walk 3 meters as quickly and safely as possible, cross a lined marked on the floor, turn around, walk back and sit down while holding a cup filled with water
Activities-Specific Confidence Scale | Baseline, Week 4, and Week 8
  16 item measure, scored from 0 to 100. Higher scores reflect great confidence of task
CNS Vital Signs - Psychomotor Speed Domain | Baseline, Week 4, and Week 8
  In-office neurocognitive test that is a non-invasive clinical procedure designed to efficiently and objectively assess a broad spectrum of brain function performance or domains under challenge. Finger tapping test and symbol digit coding will be aggregated to arrive at one reported value representing the psychomotor speed domain. Above average domain scores indicate a standard score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-109 or PR 25-74, indicating normal function. Low Average is a SS 80-89 or PR 9-24 indicating a slight deficit or impairment. Below Average is a SS 70-79 or PR 2-8, indicating a moderate level of deficit or impairment. Very Low is a SS less than 70 or a PR less than 2, indicating a deficit and impairment.
CNS Vital Signs - Executive Functioning Domain | Baseline, Week 4, and Week 8
  In-office neurocognitive test that is a non-invasive clinical procedure designed to efficiently and objectively assess a broad spectrum of brain function performance or domains under challenge. Shifting attention score will represent the executive functioning domain. Above average domain scores indicate a standard score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-109 or PR 25-74, indicating normal function. Low Average is a SS 80-89 or PR 9-24 indicating a slight deficit or impairment. Below Average is a SS 70-79 or PR 2-8, indicating a moderate level of deficit or impairment. Very Low is a SS less than 70 or a PR less than 2, indicating a deficit and impairment.
CNS Vital Signs - Reaction Time Domain | Baseline, Week 4, and Week 8
  In-office neurocognitive test that is a non-invasive clinical procedure designed to efficiently and objectively assess a broad spectrum of brain function performance or domains under challenge. Stroop test score will represent the reaction time domain. Above average domain scores indicate a standard score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-109 or PR 25-74, indicating normal function. Low Average is a SS 80-89 or PR 9-24 indicating a slight deficit or impairment. Below Average is a SS 70-79 or PR 2-8, indicating a moderate level of deficit or impairment. Very Low is a SS less than 70 or a PR less than 2, indicating a deficit and impairment.
CNS Vital Signs - Cognitive Flexibility Domain | Baseline, Week 4, and Week 8
  In-office neurocognitive test that is a non-invasive clinical procedure designed to efficiently and objectively assess a broad spectrum of brain function performance or domains under challenge. Shifting attention test and Stroop test scores will be aggregated to arrive at one reported value representing the cognitive flexibility domain. Above average domain scores indicate a standard score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-109 or PR 25-74, indicating normal function. Low Average is a SS 80-89 or PR 9-24 indicating a slight deficit or impairment. Below Average is a SS 70-79 or PR 2-8, indicating a moderate level of deficit or impairment. Very Low is a SS less than 70 or a PR less than 2, indicating a deficit and impairment.
Physical Activity Enjoyment Scale | Week 1, Week 2, Week 3, and Week 4
  scale of participant enjoyment in the moment. 7-point bipolar rating scale, eleven items are reverse scored. Higher total score reflect greater levels of enjoyment
Global Impression of Change | Week 1, Week 2, Week 3, Week 4, and Week 8
  9 point Likert scale. Higher positive score reflects great improvement
Heart Rate | Baseline, Week 1, Week 2, Week 3, Week 4, and Week 8
  heart rate beats per minute
Blood Pressure | Baseline, Week 1, Week 2, Week 3, Week 4, and Week 8
  systolic and diastolic, mm/Hg

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States